CLINICAL TRIAL: NCT06990763
Title: Clinical and Molecular Mechanism Study of Remimazolam Regulating the N/OFQ-inflammation-immune Axis to Optimize the Effect of General Anesthesia in Gynecological Surgery
Brief Title: Network Pharmacology Was Applied to Explore the Mechanism of Remimazolam Applied in General Anesthesia for Gynecological Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, professor, Second Hospital of Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hanyi20250408
Record Dates: First submitted 2025-04-20; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Gynecological Disease
Keywords: remimazolam; propofol; gynecological disease
MeSH Terms: conditions — Genital Diseases, Female | interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): Remimazolam was used for anesthesia induction and maintenance
  Interventions: Drug: Remimazolam
- Propofol group (Active Comparator): Anesthesia induction and maintenance were carried out using propofol
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam, sufentanil and rocuronium were used during induction, and remimazolam and refentanil were used during maintenance
  Arms: Remimazolam group
Drug: propofol — Propofol, sufentanil and rocuronium were used during induction, and propofol and remifentanil were used during maintenance
  Arms: Propofol group

SUMMARY:
To explore the related mechanisms by which remimazolam regulates hemodynamic stability, inflammatory factors and the immune system in patients undergoing general anesthesia for gynecological surgeries.

DETAILED DESCRIPTION:
①Clinical effect evaluation of remimazolam

1. Compare the hemodynamic stability (heart rate, mean arterial pressure, blood oxygen saturation), anesthesia efficiency (induction time, recovery time), and safety (incidence of adverse reactions such as hypotension, hypoxemia, and injection pain) of remimazolam alone, propofol alone, and their combination in general anesthesia for gynecological surgeries.
2. Clarify the optimal dose range of remimazolam and its synergistic effect with propofol, and optimize the anesthetic medication regimen.

   * The regulatory effect of remimazolam on the inflammation-immune axis and oxidative stress Detect the dynamic changes of serum inflammatory factors (IL-6, IL-10, TNF-α), immune indicators (CD3+, CD4+, CD4+/CD8+) and oxidative stress markers (SOD, MDA) of patients before and after the operation, and analyze the regulatory effect of remimazolam on the above indicators.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or their family members sign the informed consent form
2. Age: 18-64 years old, BMI: 18-30kg/m2
3. ASA Grade Ⅰ or Ⅱ
4. Patients undergoing gynecological surgeries (laparoscopic total hysterectomy, adnexectomy and myomectomy)

Exclusion Criteria:

1. People who are allergic to remimazolam or benzodiazepinesThyroid disease
2. Long-term use of benzodiazepines
3. Pregnancy or lactation
4. Have a history of drug abuse or alcoholism
5. Patients with contraindications for surgery
6. Patients with hypertension (clinically diagnosed with hypertension) and patients with coronary heart disease (with typical angina pectoris symptoms and excluding aortic valve lesions, with a clear history of old myocardial infarction, with a clear history of acute myocardial infarction, and CAG finding coronary artery stenosis greater than or equal to 70%)
7. Patients with arrhythmia, heart failure, renal failure, and those who have recently taken cardiovascular active drugs
8. Endocrine disorders such as hyperthyroidism and pheochromocytoma that may affect the hemodynamic level of the body
9. Patients with ketoacidosis and lactic acidosis
10. Abnormal liver function, ALT> three times the upper limit of the normal value;
11. Renal failure (serum creatinine >3mg/dl or creatinine clearance rate <30ml/min)
12. Patients who have been using sedatives or antidepressants for a long time, or have a history of alcohol abuse or drug dependence
13. Asthma or reactive airway diseases
14. Combined with underlying cognitive function abnormalities
15. Exclusion criteria for research subjects
16. Those who were mistakenly included without meeting the inclusion criteria
17. Those who experienced adverse events such as shock, severe hypotension and severe arrhythmia during the operation

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Levels of serum N/OFQ, IL-6, STAT3 | perioperatively/periprocedurally

SECONDARY OUTCOMES:
Heart rate | during the surgery
mean arterial pressure | during the surgery

CONTACTS AND LOCATIONS:
Overall Officials: yi Han, Study Director — Second Hospital of Shanxi Medical University

IPD SHARING:
Plan to Share IPD: No